CLINICAL TRIAL: NCT03247374
Title: Bio-feedback Treatment Versus Standard Treatment for Dysphagic Post-stroke Patients: a Randomized Controlled Trial
Brief Title: Bio-feedback Treatment for Dysphagic Post-stroke Patients
Acronym: BIO_DYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Sara Nordio, Speech and language therapist, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017.12 - BioDis
Record Dates: First submitted 2017-07-20; First posted 2017-08-11 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Dysphagia, Late Effect of Stroke; Deglutition Disorders
Keywords: rehabilitation; treatment; biofeedback; bio-feedback; dysphagia; swallowing disorders; post-stroke; deglutition disorders
MeSH Terms: conditions — Deglutition Disorders | interventions — Language Therapy

STUDY DESIGN:
Intervention Model Description: simple randomization into two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "ProComp5 Infiniti" Biofeedback (Experimental): Each participant will attend 5 sessions per week for a total duration of 5 weeks. The duration of each session will take 1 hour, including bio-feedback preparation. At the beginning of the bio-feedback session, a surface electrode will be applied to the mylohyoid muscle. The patient will be required to swallow at a given time, with food bolus if possible, and perform maneuvers that favour swallowing strength and efficacy: effortful swallow, supraglottic swallow, and "Masako" maneuver, the first two with bolus administration, if possible. The experimental group will perform this training for 45 minutes, plus they will receive a verbal feedback from the speech and language therapist.
  Interventions: Device: "ProComp5 Infiniti" Biofeedback
- Standard Speech and Language Therapy (Active Comparator): Each participant will attend 5 sessions per week for a total duration of 5 weeks. The patient will be required to swallow at a given time, with food bolus if possible, and perform maneuvers that favour swallowing strength and efficacy: effortful swallow, supraglottic swallow, and "Masako" maneuver, the first two with bolus administration, if possible. The control group will attend this training for 45 minutes, receiving verbal feedback from the speech and language therapist.
  Interventions: Other: Standard Speech and Language Therapy

INTERVENTIONS:
Device: "ProComp5 Infiniti" Biofeedback — Each participant will attend 5 sessions per week for a total duration of 5 weeks. At the beginning of the bio-feedback session, a surface electrode will be applied to the mylohyoid muscle. The computer will produce visual feedback of the muscular activity on the screen. The patient will be required to swallow at a given time, with food bolus if possible, and perform maneuvers that favour swallowing strength and efficacy: they are requested to do classical maneuvers that favour swallowing efficacy that is effortful swallow, supraglottic swallow, and "Masako" maneuver. The experimental group will perform this training for 45 minutes.
  Arms: "ProComp5 Infiniti" Biofeedback
Other: Standard Speech and Language Therapy — Each participant will attend 5 sessions per week for a total duration of 5 weeks. The patient will be required to swallow at a given time, with food bolus if possible, and perform maneuvers that favour swallowing strength and efficacy receiving verbal feedback from the speech and language therapist. They are requested to do classical maneuvers that favour swallowing efficacy that is effortful swallow, supraglottic swallow, and "Masako" maneuver. The control group will perform this training for 45 minutes.
  Arms: Standard Speech and Language Therapy

SUMMARY:
The primary purpose of the study is to evaluate whether the effect of bio-feedback dysphagia treatment is more effective than a control treatment in post-stroke patients.

This study will be a randomized, single-blind controlled pilot study. The investigators intend to recruit 40 patients who have suffered a stroke and have dysphagia. Twenty patients will undergo training with bio-feedback (experimental group) and the other 20 patients will undergo standard training, using only verbal feedback rather than visual feedback (control group).

The authors hypothesize that in the control group the efficacy of the treatment will be lower in the absence of immediate visual feedback of strength and coordination of the swallowing act.

DETAILED DESCRIPTION:
The procedure is divided into 5 parts:

* Clinical and instrumental evaluation (fibroendoscopy) of swallowing functions before the treatment;
* 25 sessions with bio feedback treatment or 25 sessions of control treatment;
* Clinical and instrumental evaluation (fibroendoscopy) of swallowing functions after the training;
* Clinical and instrumental evaluation (fibroendoscopy) of swallowing functions after 3 months.

Each participant will attend 5 sessions per week for a total duration of 5 weeks. The duration of each session will take 1 hour, including bio-feedback preparation that will take about 10 minutes for assembly and 5 minutes for removal. At the beginning of the bio-feedback session, a surface electrode will be applied to the mylohyoid muscle. The computer will analyze the electromyographic signal of the patient in real time and will produce visual feedback of the muscular activity on the screen. The patient will be required to swallow at a given time, with food bolus if possible, and perform maneuvers that favor swallowing strength and efficacy.

During the first session, participant will be instructed to use the tool before starting the training phase. Patients of both groups will participate in similar sessions, with classical maneuvers favoring swallowing efficacy that is effortful swallow, supraglottic swallow, and "Masako" maneuver, the first two with bolus administration, if possible. The experimental group will perform this training for 45 minutes with the support of visualization of muscle activity on the screen (biofeedback), while the control group will attend the same training for 45 minutes, but receiving verbal feedback from the speech and language therapist.

Data analysis

On the measures collected, a descriptive statistical analysis and distribution will be studied. Initial instrumental and clinical data from FOIS scale (The Functional Oral Intake Scale), PAS (Penetration-Aspiration Scale), Pooling Score (Farneti et al.); Cranial nerves test will be analyzed using parametric (t-test) and non-parametric (Wilcoxon test) tests with a p-value considered significant if <0.05, while longitudinal variations will be analyzed using ANOVA for repeated measurements. In addition, the effect size (Cohen's d) of the difference between the instrumental and clinical evaluation scales average before and after training in both groups will be calculated. This will allow to have an estimate of training effectiveness to perform a power study and plan a wider experimental study for validating the method.

ELIGIBILITY:
Inclusion Criteria:

* first stroke injury
* single lesion
* onset from more than six weeks
* presence of dysphagia (Dysphagia Outcome and Severity Scale ≥ 4)
* good comprehension ( not below PT 53 in Token Test)
* good eyesight and hearing, or adequately corrected

Exclusion Criteria:

* All the elements that hinder a good recording of the electromyographic signal (for instance a cutaneous infection, a wound or a dermatitis in the submandibular area);
* Severe concomitant illnesses (fever, infections, metabolic problems, serious cardiac insufficiency) that can influence patient's collaboration;
* Serious dystonia or unintentional movements
* presence of disorders of consciousness;
* encephalopathy due to multiple infarcts;
* inability to sustain the experimental treatment;
* other neurological diseases (for example Parkinson disease);

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Functional Oral Intake Scale (FOIS) | Baseline , 4 weeks , finally after 3 months from the end of treatment
  It is a 7-point scale developed to systematically rate the functional severity of dysphagia

SECONDARY OUTCOMES:
Change in Pooling Score (P-score) | Baseline , 4 weeks , finally after 3 months from the end of treatment
  The scale is used during clinical endoscopic evaluation to evaluate severity of swallowing disorder, considering excess residue in the pharynx and larynx.The score (minimum 4 - maximum 11) is obtained by the sum of the scores given to the site of the bolus, the amount and ability to control residue/bolus pooling, the latter assessed on the basis of cough, raclage, number of dry voluntary or reflex swallowing acts.
Change in Penetration-Aspiration Scale (PAS) | Baseline , 4 weeks , finally after 3 months from the end of treatment
  It is a 8-point scale used during endoscopic evaluation that describes and measures the severity of airway invasion during swallowing.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Nordio, Principal Investigator — IRCCS San Camillo
Locations (1):
- Sara Nordio, Venice-Lido, Italy